CLINICAL TRIAL: NCT01184261
Title: Integrated Intervention for Cigarette Smoking and Binge Drinking for Young Adults
Brief Title: Integrated Behavioral Intervention for Cigarette Smoking and Binge Drinking in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Principal Investigator, Steven Ames, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-000432; NCI-2010-01881
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: for Cigarette Smoking and Binge Drinking Cessation
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients attend behavioral sessions for smoking and binge drinking cessation over 30 minutes once weekly in weeks 1-6.
  Interventions: Behavioral: behavioral intervention
- Arm II (Experimental): Patients attend behavioral sessions for smoking cessation over 30 minutes once weekly in weeks 1-6.
  Interventions: Behavioral: behavioral intervention

INTERVENTIONS:
Behavioral: behavioral intervention — 8 session behavioral intervention.
  Other Names: Behavior or Life Style Modifications; Behavior Therapy; Behavioral Modification; Behavioral Therapy; Behavioral Treatment

SUMMARY:
RATIONALE: Nicotine patches and behavioral therapy may help reduce cigarette smoking and binge drinking in young adults. PURPOSE: This randomized clinical trial studies nicotine patches with or without behavioral therapy in reducing cigarette smoking and binge drinking in young adults.

DETAILED DESCRIPTION:
OBJECTIVES: I. To evaluate the efficacy of Integrated Intervention that targets both cigarette smoking and binge drinking on the cigarette smoking behavior of young adult smokers at 6-month follow-up. II. To evaluate the efficacy of Integrated Intervention that targets both cigarette smoking and binge drinking on binge drinking behavior of young adult smokers. III. Examine the effect of Integrated Intervention on several possible mediators of change corresponding to mechanisms that have been proposed to account for the relationship between cigarette smoking and alcohol use. These mediators include cravings to smoke, perceived similarity to the typical smoker, and self-efficacy for smoking abstinence. OUTLINE: Patients are randomized to 1 of 2 treatment arms.All patients receive nicotine patch therapy in weeks 4-11. ARM I: Patients attend behavioral sessions for smoking and binge drinking cessation over 30 minutes once weekly in weeks 1-6. ARM II: Patients attend behavioral sessions for smoking cessation over 30 minutes once weekly in weeks 1-6.After completion of study treatment, patients are followed up at weeks 12, 16, 20, and 24.

ELIGIBILITY:
Inclusion Criteria: - Smoked an average of >= 10 or more cigarettes per day during the past 6 months - Binge drank on an average of >= 2 occasions per month during the past 3 months - Able to participate fully in all aspects of the intervention and keep all scheduled appointments - Willing to participate in 6 months of follow-up - Willing to stop smoking and use nicotine patch therapy - Willing to refrain from participating in additional smoking interventions for the duration of the study - Provide written informed consent Exclusion Criteria: - Current (past 90 days) alcohol dependence as assessed by the Structured Clinical Interview for DSM-IV Axis I Disorders, Alcohol Dependence Module - Current (past 12 months) non-nicotine or alcohol drug dependence as assessed by a Drug Abuse Screening Test-20 score of >= 6 - Current elevation of depressive symptoms (past 2 weeks) that would be indicative of clinical depression as assessed by a Beck Depression Inventory-II score of >= 20 - Current use (past 30 days) of nicotine containing medication or frequent use (> 10 occasions per month) of tobacco products other than cigarettes - Current use (past 30 days) of any other smoking cessation treatment involving behavioral or pharmacological interventions - Any medical condition that would preclude use of the nicotine patch including current unstable angina, recent history (past 30 days) of myocardial infarction or stroke, history of severe skin allergies, or evidence of severe chronic dermatosis - Currently pregnant or breast feeding, or likely to become pregnant during the nicotine patch phase

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2010-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Biochemically-confirmed 7-day point prevalence tobacco abstinence | At week 24

SECONDARY OUTCOMES:
Effect of the integrated intervention on binge drinking | At week 24
Possible mediators of the intervention | At week 24

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ames, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States